CLINICAL TRIAL: NCT01505140
Title: Benefits of Walnuts for Male Reproductive Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 445246WR77518
Record Dates: First submitted 2011-12-31; First posted 2012-01-06 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Infertility; Nutrition Disorders
Keywords: Andrology; Fertility; Reproduction; Diet; Nutritional Sciences; Fatty Acids; Antioxidants; Body weight changes
MeSH Terms: conditions — Infertility; Nutrition Disorders; Body Weight Changes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Western style diet (No Intervention): Participants will consume their usual Western style diet avoiding tree nuts
- Whole walnuts (Experimental): Participants will consume usual Western style diet adding 75 gm whole walnuts per day
  Interventions: Other: Whole walnuts

INTERVENTIONS:
Other: Whole walnuts — 75 gm whole walnuts per day will be consumed with usual Western style diet
  Arms: Whole walnuts

SUMMARY:
Walnuts as a whole food contain polyunsaturated fatty acids, anti-oxidants, and other nutrients essential to sperm development and function. This randomized controlled trial sought to determine if a Western style diet supplemented with walnuts would improve sperm quality as a predictor of male fertility.

DETAILED DESCRIPTION:
A vast research base on human sperm shows the following to be critical for normal sperm development and function: Polyunsaturated fatty acids provide fluidity to sperm membranes allowing sperm to swim, fuse with ova, and support key cellular functions. Antioxidants protect sperm from reactive oxygen species generated during normal physiologic processes or white blood cells that infiltrate into seminal fluid and injure membranes and fragment sperm DNA. Selenium is critical in the form of anti-oxidant selenoproteins protecting developing sperm in the testes and later selenium in the epididymis participates in cell shape for motility. Folate, in a recent study, was associated with decreased aneuploidy (abnormal number of chromosomes)in sperm. Deficiency in any of these factors - lipids, antioxidants, selenium, or folate could manifest as poor semen quality and sub-fertility.

Walnuts provide a rich dietary source of each of the critical factors discussed above. Walnuts contain beneficial lipids, antioxidants, selenium, and folate. Walnuts, as a natural whole food source, may be preferential to commercial supplements and, as a plant source of nutrients, leave a positive green footprint on the planet.

Hypothesis The investigators hypothesize that diets enriched in walnuts will improve semen quality. Semen quality is a predictive marker for male infertility and sub-fertility, thus, the overall goal is to determine if dietary intake of walnuts will benefit male reproductive health.

A randomized, controlled intervention will be used to study the effects of walnut supplementation on semen quality measures in young men (ages 21 to 35) eating Western diets. Participants will be enrolled from the West Los Angeles area (n=120). Men will be randomly assigned to consume 3 oz of walnuts per day as part of their usual diet or to continue their habitual diet but avoid nuts. Each will follow the assigned diet for three months to cover one complete cycle of spermatogenesis.

The specific aims of the study are to:

1. Establish at baseline: habitual diet; serum omega-3 to omega-6 ratio, serum selenium and folate; semen quality (sperm count, motility, morphology) and sperm DNA integrity (COMET assay); sperm aneuploidy; and semen anti-oxidant levels
2. Randomly assign men to habitual diet plus 3 oz walnuts per day or usual diet without nuts for three months monitored by six telephone 24 hour dietary recalls
3. Compare intervention and control groups at three months on blood and semen measures
4. Compare blood and semen measures within man between baseline and three months.

ELIGIBILITY:
Inclusion Criteria: Males

1. Age 21 to 35 years
2. Residence is in West Los Angeles for the next three months
3. Non-smoker
4. Free from chronic diseases requiring medications
5. Free from nut allergies or nut intolerance
6. Not taking anti-oxidant supplements

Exclusion Criteria:

1. Outside the age range of 21 to 35 years
2. Residence outside West Los Angeles area prohibiting two trips to the clinical research laboratory
3. Current smoker
4. Taking medications for chronic disease
5. Nut allergies or nut intolerance
6. Taking anti-oxidant supplements -

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
change from baseline in semen quality at 12 weeks | change from baseline at 12 weeks
  semen quality is measured as sperm count, motility, vitality, morphology, DNA integrity
change from baseline in serum fatty acids at 12 weeks | change from baseline at 12 weeks
change from baseline in serum selenium at 12 weeks | change from baseline at 12 weeks
change from baseline in serum folate at 12 weeks | change from baseline at 12 weeks
change from baseline in serum zinc at 12 weeks | change from baseline at 12 weeks

SECONDARY OUTCOMES:
change from baseline in body weight pounds at 12 weeks | change from baseline at 12 weeks
change from baseline in nutrient intake at 12 weeks | change from baseline at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendie A Robbins, RN, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Robbins WA, Xun L, FitzGerald LZ, Esguerra S, Henning SM, Carpenter CL. Walnuts improve semen quality in men consuming a Western-style diet: randomized control dietary intervention trial. Biol Reprod. 2012 Oct 25;87(4):101. doi: 10.1095/biolreprod.112.101634. Print 2012 Oct. PMID 22895856